CLINICAL TRIAL: NCT05594199
Title: Development and Evaluation Of A Virtual Smoking Cessation Program - A Pilot Study
Brief Title: Feasibility of a Virtual Smoking Cessation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jean Wong, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-5475
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Smoking; Smoking Cessation; Smoking Reduction; Perioperative/Postoperative Complications; Fractures, Bone
Keywords: Smoking; Smoking Cessation; Electronic Mail; Virtual Program; Fracture; Surgery; Perioperative
MeSH Terms: conditions — Smoking; Smoking Cessation; Smoking Reduction; Postoperative Complications; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm: Virtual Group (Experimental): The intervention will involve participating in the study's virtual smoking cessation program. This program consists of 2 components: an e-learning module and a tailored email messaging program based on the participant's motivation to quit smoking and their Fagerstrom test for nicotine dependence score.
  Interventions: Behavioral: Virtual Smoking Cessation Program
- Control Arm: Standard Care (No Intervention): This arm will receive standard care which may or may not include brief advice to quit smoking from any of the healthcare providers.
  Providing smoking cessation intervention is not mandatory in standard care and may not be provided.

INTERVENTIONS:
Behavioral: Virtual Smoking Cessation Program — This program consists of an e-learning smoking cessation education module and a tailored email messaging program.
  The e-learning module addresses the potential health benefits to quitting smoking regarding surgery or recovering from a fracture. In addition, it provides information on getting support through the process of quitting smoking based on the individual's level of smoking dependence.
  Email frequency and content will vary based on the participant's score and level of motivation. Information will include the risks associated with smoking before surgery or how quitting smoking can improve recovery from a fracture injury. Additional information includes the benefits of quitting smoking and developing coping strategies during a quit attempt. Motivational emails and references to free resources for additional smoking cessation support will also be provided.
  Arms: Intervention Arm: Virtual Group

SUMMARY:
The goal of this pilot study of a clinical trial is to learn about the acceptability and feasibility of a virtual smoking cessation program in both the perioperative and fracture clinic settings. The main questions this study aims to answer are:

* The number of people that participate in the virtual smoking cessation program
* The acceptability of the number, length, content, and delivery of the email messages provided by the program.

Participants will be asked to subscribe to our virtual intervention which will include:

* A smoking cessation e-learning module component to provide education on the risks of smoking in the surgical or fracture clinic setting, and
* An emailing program component that will provide tailored email messages over a 30-45 day period depending on a patient's Fagerstrom test for nicotine dependence score and motivation to quit smoking.

Researchers will also compare the virtual smoking cessation program to standard care to see if there are any differences shown between both groups in the Fagerstrom test for nicotine dependence scores, number of cigarettes smoked, number of quit attempts, complication rates, and re-admission rates at the 7 day and 30 day time points.

DETAILED DESCRIPTION:
Smoking is the most preventable cause of disease and premature death in Canada. In this pilot study our aim is to determine whether a virtual perioperative program, using automated emails, for smoking cessation is feasible and acceptable for increasing abstinence from smoking, compared to the usual care in patients undergoing surgery or with an acute traumatic fracture. Patients that present to the preoperative clinic or fracture clinic will be recruited for this trial. This feasibility study will be followed by the proposed randomized control trial to identify whether our planned study procedures are acceptable to surgical patients.

Both components of the virtual smoking cessation program (Smoking cessation e-learning modules and Virtual Program Evaluation) will be more personalized to the patient as the patient's nicotine dependence will determine the tailored information that will be provided in the e-learning module and the email messages. Study procedures and components of the virtual smoking cessation program will be modified for clinical use and future research based on the feedback from this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Daily or non-daily smoker
* Self-reported smokers who have smoked cigarettes within the past 30 days
* Must be a patient at Toronto Western Hospital or Women's College Hospital who is:

  * Scheduled for an elective surgical procedure that will occur at least 48 hours after recruitment OR
  * Visiting the fracture clinic (UHN) within and including 14 days from the initial date of injury or operation
* Must have a working e-mail address

Exclusion Criteria:

* Patients who have already quit smoking for more than 30 days,
* Patients who cannot read and understand English,
* Patients who have any form of cognitive impairment,
* Patients who do not have a telephone (for follow-up).
* Currently on pharmacological therapy for smoking cessation
* Drug or alcohol abuse or dependence within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Trial feasibility - Recruitment | Surgery: 30 days after surgery; Fracture Clinic: 30 days
  Feasibility as assessed by recruitment rate. This will be assessed as the proportion of participants who agree to participate compared to the number of patients who had met the inclusion/exclusion criteria and were approached to participate in the study.
  The demographics of those who declined to participate or dropped out of the virtual program will be assessed for trends within the population who do not wish to participate in the virtual smoking cessation program
Trial feasibility - Acceptability of the email message program component | Surgery: 30 Days after surgery; Fracture Clinic: 30 days after study recruitment
  Patients will be asked to evaluate the email program and messages provided during their participation in the virtual program through a questionnaire that will evaluate the frequency, length, content, delivery, and duration of the email message component using a 5-point Likert scale.
Trial feasibility - Acceptability of e-learning module program component | Surgery: Before surgery; Fracture Clinic: Day 7 after study recruitment
  Patients will be asked to evaluate the e-learning module once they completed it. A survey will be administered to evaluate the content and comprehension of the e-learning module using a 5-point Likert scale.
Trial feasibility - EPIC patient portal usage | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  The feasibility of delivering this virtual program through the patient portal will be assessed by the proportion of study participants who have self-reported patient portal use compared to the total number of study participants.
Trial feasibility - Retention | Surgery: 30 days after surgery; Fracture Clinic: 30 days
  Feasibility as assessed by the retention rates. This will be defined as the proportion of program participants completing the study at the final follow-up compared to the participants enrolled.
  Reasons for withdrawal will also be recorded to assess any trends that occur among participants who drop out.

SECONDARY OUTCOMES:
Module Education | At time of recruitment, and after module completion (Surgery: Before surgery; Fracture Clinic: Day 7 after study recruitment)
  The effectiveness of the virtual program's e-learning module component will be assessed by a survey that will evaluate the patient's understanding of the risks of smoking before/after surgery and while recovering from a fracture using a 5-point Likert scale.
Cigarettes smoked | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  The number of cigarettes smoked per day.
Quit attempts | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  The number of quit attempts made since study recruitment.
  A quit attempt will be defined by a patient making a serious, conscious attempt to completely abstain from cigarette smoking and has abstained from smoking for at least 24 hours.
Nicotine Dependence | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  Nicotine dependence will be assessed using the Fagerström test for nicotine dependence, which is a standard instrument for assessing the intensity of physical addiction to nicotine.
Stage of change | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  Stage of Change will be assessed using Prochaska and DiClemente's Stages of Change Model, a transtheoretical model of change that proposes a series of stages through which smokers move as they successfully change their smoking habit.
Self or assisted quit attempt | Surgery: (i)Day of recruitment, (ii)Day of Surgery, (iii) 7 day follow-up, (iv) 30 day follow-up; Fracture Clinic: (i)Day of recruitment, (ii)7 day follow-up, (iii) 14 day follow-up, (iv) 30 day follow-up
  Participants will be asked to report whether they are currently going through a self-quit attempt or a quit attempt assisted by a health care professional
Complications/Adverse Events | Surgery: 30 days after surgery; Fracture Clinic: 30 days after study recruitment
  Complications/adverse events regarding the patient's surgery or recovery from fracture will be obtained from the patient's electronic health record.
Readmission | Surgery: 30 days after surgery; Fracture Clinic: 30 days after study recruitment
  The number of readmissions to the hospital will be obtained from the patient's electronic health record.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Graham AL, Carpenter KM, Cha S, Cole S, Jacobs MA, Raskob M, Cole-Lewis H. Systematic review and meta-analysis of Internet interventions for smoking cessation among adults. Subst Abuse Rehabil. 2016 May 18;7:55-69. doi: 10.2147/SAR.S101660. eCollection 2016. PMID 27274333
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Andersen T, Christensen FB, Laursen M, Hoy K, Hansen ES, Bunger C. Smoking as a predictor of negative outcome in lumbar spinal fusion. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2623-8. doi: 10.1097/00007632-200112010-00018. PMID 11725245
- [Background] Mills E, Eyawo O, Lockhart I, Kelly S, Wu P, Ebbert JO. Smoking cessation reduces postoperative complications: a systematic review and meta-analysis. Am J Med. 2011 Feb;124(2):144-154.e8. doi: 10.1016/j.amjmed.2010.09.013. PMID 21295194
- [Background] Myers K, Hajek P, Hinds C, McRobbie H. Stopping smoking shortly before surgery and postoperative complications: a systematic review and meta-analysis. Arch Intern Med. 2011 Jun 13;171(11):983-9. doi: 10.1001/archinternmed.2011.97. Epub 2011 Mar 14. PMID 21403009